CLINICAL TRIAL: NCT04499846
Title: Can Educational Intervention Targeting Statin Therapy Improve Compliance in Diabetic Patients
Brief Title: Educational Intervention Targeting Statin Therapy and Compliance in Diabetic Patients
Acronym: STADIA
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0096; 2020-A00402-37 (Other: IDRCB)
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Type II Diabetes
Keywords: Diabetes; Compliance; Statin; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients following education: Patients will followed an educational intervention about physiopathology of diabetes and mechanisms of action of statins. A questionnaire will allow to measure compliance to the treatment.
  Interventions: Other: Therapeutic education

INTERVENTIONS:
Other: Therapeutic education — Patients will follow a therapeutic education in order to inform them about the mechanism of action of statins. After this intervention a questionnaire will use to measure compliance.

SUMMARY:
The objective of the study is to measure changes in compliance to statin therapy in patients with type 2 diabetes after an educational intervention. This intervention is part of the therapeutic education of the diabetic patient, carried out throughout the follow-up of his/her diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Type 2 diabetes
* Following treatment with statins
* Hospitalization in the diabetes day hospitals of the Saint Philibert or Saint Vincent Hospitals (Lille, France).
* Ability to answer the Girerd test in both interviews (in the individual interview and by phone)
* Patient informed to participate in the study
* Signed patient's consent.

Exclusion Criteria:

* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients hospitalized in the diabetes day hospitals of the Saint Philibert or Saint-Vincent hospitals (Lille, France)
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Compliance rate to the statin treatment | 3 months
  Compliance is estimated with the compliance evaluation Test of Girerd based on a score from 0 to 6. Six questions are asked to the patient.
  For the interpretation of the test:
  Total YES = 0, Score = 0: Good compliance Total YES = 1 or 2, Score = 1 or 2: Minimal compliance Total YES ≥ 3, Score ≥ 3: Poor compliance Lack of completion of the questionnaire is considered as "poor compliance".

SECONDARY OUTCOMES:
Compliance rate to the statin treatment according to schedule of drug intake | 3 months
  Compliance is estimated with the compliance evaluation Test of Girerd based on a score from 0 to 6. Six questions are asked to the patient.
  For the interpretation of the test:
  Total YES = 0, Score = 0: Good compliance Total YES = 1 or 2, Score = 1 or 2: Minimal compliance Total YES ≥ 3, Score ≥ 3: Poor compliance Lack of completion of the questionnaire is considered as "poor compliance".
Compliance rate to the statin treatment according to treatment duration. | 3 months
  Compliance is estimated with the compliance evaluation Test of Girerd based on a score from 0 to 6. Six questions are asked to the patient.
  For the interpretation of the test:
  Total YES = 0, Score = 0: Good compliance Total YES = 1 or 2, Score = 1 or 2: Minimal compliance Total YES ≥ 3, Score ≥ 3: Poor compliance Lack of completion of the questionnaire is considered as "poor compliance".

CONTACTS AND LOCATIONS:
Overall Officials: François Delecourt, MD, Principal Investigator — GHICL
Locations (1):
- Hôpital Saint-philibert, Lomme, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No